CLINICAL TRIAL: NCT05512598
Title: Multi-centre, Open-label, Single-arm, Phase Ib Study to Evaluate the Safety, Pharmacokinetics, and Efficacy of a Single Dose of HB0034 in Patients Acute Generalized Pustular Psoriasis (GPP) Flare
Brief Title: HB0034 in Patients With Generalized Pustular Psoriasis (GPP)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Huaota Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HB0034-02
Record Dates: First submitted 2022-08-22; First posted 2022-08-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Generalized Pustular Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HB0034 (Experimental): Recombinant Humanized Anti-IL-36R Monoclonal antibody
  Interventions: Drug: HB0034

INTERVENTIONS:
Drug: HB0034 — HB0034, a single dose
  Other Names: HB0034, a recombinant humanized anti-IL-36R IgG1 monoclonal antibody

SUMMARY:
This is a study to evaluate the safety, tolerability, pharmacokinetics, and efficacy of HB0034 in adult patients with generalized pustular psoriasis (GPP ).

DETAILED DESCRIPTION:
This is an open-label, multicenter, phase Ib exploratory study to evaluate the safety, tolerability, pharmacokinetics, and efficacy of HB0034 in adult patients presenting moderate-severe generalized pustular psoriasis (GPP ) flare.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, aged 18 to 75 years at screening
* A known and documented history of Generalized Pustular Psoriasis diagnosed with ERASPEN criteria
* Presenting with a moderate-severe flare of Generalized Pustular Psoriasis (GPP)
* Patients must be able to understand and sign a written informed consent document and complete study-related procedures and questionnaires.

Exclusion Criteria:

* Immediate life-threatening flare of Generalized Pustular Psoriasis or requiring intensive care treatment, according, to the judgment of the investigator. Life-threatening complications mainly include but are not limited to, cardiovascular/cytokine-driven shock, pulmonary distress
* History of clinically significant opportunistic infection (e.g., invasive candidiasis or pneumocystis pneumonia)
* Pregnant or Breasting feeding subject. Women with a positive pregnancy test.
* Ongoing use of prohibited psoriasis treatments
* Further exclusions criteria apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-11-06 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Number of patients with drug related adverse events | 90 days
  An AE is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of investigational drug

SECONDARY OUTCOMES:
Proportion of Patients achieved GPPAG pustular 0/1 (pustular cleared or almost cleared) | 12 weeks
  efficacy outcome of investigational drug
Cmax | 12 weeks
  The maximum measured concentration of the analysis in plasma
AUC0-infinity | 12 weeks
  The area under the concentration-time curve of the analysis in plasma over the time interval from 0 extrapolated to infinity

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Furen, Doc., Principal Investigator — Shandong Provincial Dermatology Hospital
Locations (1):
- Dermatology Hospital of Shandong First Medical University, Shandong, Shandong, China

IPD SHARING:
Plan to Share IPD: No